CLINICAL TRIAL: NCT02888327
Title: A Phase-1, Open-label, Four Group, Fixed-Sequence Study to Evaluate the Effect of AL-794 on the Pharmacokinetics of Oseltamivir, JNJ-63623872, and Probes for P-glycoprotein, CYP3A and OATP1B1 in Healthy Volunteers
Brief Title: A Drug-Drug Interaction Study to Evaluate the Effect of AL-794 on the Pharmacokinetics of Oseltamivir and JNJ-63623872
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL-794-802
Record Dates: First submitted 2016-08-19; First posted 2016-09-05 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Influenza in Humans
MeSH Terms: conditions — Influenza, Human | interventions — sfericase; Oseltamivir; Digoxin; Midazolam; pitavastatin; pimodivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Oseltamivir and AL-794 (Other): Oseltamivir alone and with AL-794 over fourteen days.
  Interventions: Drug: AL-794; Drug: Oseltamivir
- Digoxin, Midazolam, and AL-794 (Other): Single doses of Digoxin and Midazolam with and without AL-794 over seventeen days.
  Interventions: Drug: AL-794; Drug: Digoxin; Drug: Midazolam
- Pitavastatin and AL-794 (Other): Single doses of Pitavastatin with and without AL-794 over seventeen days.
  Interventions: Drug: AL-794; Drug: Pitavastatin
- JNJ-63623872 and AL-794 (Other): JNJ-63623872 alone and with AL-794 over fourteen days.
  Interventions: Drug: AL-794; Drug: JNJ-63623872

INTERVENTIONS:
Drug: AL-794
Drug: Oseltamivir
  Arms: Oseltamivir and AL-794
Drug: Digoxin
  Arms: Digoxin, Midazolam, and AL-794
Drug: Midazolam
  Arms: Digoxin, Midazolam, and AL-794
Drug: Pitavastatin
  Arms: Pitavastatin and AL-794
Drug: JNJ-63623872
  Arms: JNJ-63623872 and AL-794

SUMMARY:
This open-label, four group, fixed-sequence study will evaluate the safety and pharmacokinetic interaction of AL-794 on oseltamivir, JNJ-63623872 (formerly VX-787) and probes for P-glycoprotein, CYP3A and OATP1B1 in healthy volunteers.

DETAILED DESCRIPTION:
This open-label, four group, fixed-sequence study will evaluate the safety and pharmacokinetic interaction of AL-794 on oseltamivir, JNJ-63623872 (formerly VX-787) and probes for P-glycoprotein, CYP3A and OATP1B1 in healthy volunteers.

For each group, the study consists of an eligibility screening period, study period, and 1 follow-up visit. Groups may enroll in parallel but subjects enrolled in one group may not participate in another group.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written consent.
2. In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions and is likely to complete the study as planned.
3. Subject is in good health as deemed by the investigator, based on the findings of a medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG).
4. Male or female, 18-60 years of age.
5. Body mass index (BMI) 18-30 kg/m2, inclusive. The minimum weight is 50 kg.
6. A female subject is eligible to participate in this study if she is of non-childbearing potential (defined as females with a documented tubal ligation, bilateral oophorectomy or hysterectomy) or postmenopausal (defined as 12 months of spontaneous amenorrhea and follicle stimulating hormone level within the laboratory's reference range for postmenopausal females). A postmenopausal female receiving hormone replacement therapy who is willing to discontinue hormone therapy 28 days before study drug dosing and agrees to remain off hormone replacement therapy for the duration of the study may be eligible for study participation. Females must refrain from donating eggs (ova, oocytes) for the purposes of assisted reproduction from check-in through 6 months after dosing.
7. If male, subject is surgically sterile or practicing acceptable forms of birth control until 90 days after the end of the study. Males must agree to refrain from sperm donation from check-in through 90 days after dosing.

Exclusion Criteria:

1. Men whose female partners are pregnant or contemplating pregnancy from the date of screening until 90 days after their last dose of study drugs.
2. Clinically significant laboratory abnormalities or abnormalities which are deemed to interfere with the ability to interpret study data.
3. Creatinine clearance of less than 60 mL/min (MDRD).
4. Total bilirubin, ALT, AST, or alkaline phosphatase >1.2× upper limit of normal (documented Gilbert's permitted).
5. Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hematologic, neurologic, thyroid or any other medical illness or psychiatric disorder, as determined by the Investigator and/or Sponsor's Medical Monitor.
6. Positive screening test for influenza, hepatitis A, B, C or human immunodeficiency virus (HIV) serology.
7. Any condition that, in the opinion of the investigator, would compromise the study's objectives or the well-being of the subject or prevent the subject from meeting the study requirements.
8. Participation in an investigational drug trial or having received an investigational vaccine within 3 months or 5 half-lives (whichever is longer) prior to study medication.
9. Clinically significant abnormal ECG findings. Particularly, a history or family history of prolonged QT syndrome (eg, torsade de pointes), pre-existing sinus node disease, (incomplete) AV block, heart failure, or sudden cardiac death; or a corrected QT interval (QTcF or QTcB) >450 milliseconds for male subjects and >470 milliseconds for female subjects at the screening visit.
10. Clinically significant blood loss or elective blood donation of significant volume (ie, >500 mL) within 90 days of first dose of study drug; >1 unit of plasma within 7 days of first dose of study drug.
11. Clinically significant abnormal heart rate, respiratory rate, temperature or blood pressure values outside of the normal range, per local standards (evaluated in a semi-recumbent or recumbent position after 5 minutes of rest) which are considered clinically significant. One repeat measurement after an additional 5 minutes of rest is permitted in one visit day.
12. Evidence or current diagnosis of sleep apnea.
13. Evidence of clinically significant infection within 2 weeks prior to admission.
14. Unwilling to abstain from alcohol for at least 1 week prior to the start of dosing through the Study Completion visit.
15. History of regular alcohol intake >14 units per week of alcohol for females and >21 units per week for males (one unit is defined as 8 g alcohol) within 3 months of the screening visit.
16. History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 1 year before screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening or Day 1.
17. History of tobacco use or used nicotine-containing products within 3 months of the screening visit.
18. The subject has a positive prestudy drug screen.
19. The use of concomitant medications, including prescription, over the counter medications, herbal medications, inducers or inhibitors of CYP enzymes, glucuronidation or drug transporters (including P-glycoprotein and OATP1B1) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication is excluded, unless approved by the Sponsor's Medical Monitor. Occasional use of paracetamol, or its equivalent, is permitted.
20. Exposure to more than 4 new investigational entities within 12 months prior to the first dosing day.
21. Hypersensitivity to the active substances or to any of the excipients of AL-794, oseltamivir, JNJ-63623872, digoxin, midazolam, or pitavastatin.
22. Unwillingness or inability to comply with the study protocol for any other reason.
23. Employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator or employees of Johnson & Johnson.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2016-07-31 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for ALS-033719, ALS-033927, oseltamivir, oseltamivir carboxylate, JNJ-63623872, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on days 7, 8, and 14 for ALS-033719, ALS-033927, and JNJ-63623872
Area under plasma concentration-time curve from time 0 to dosing interval (tau) (AUC0-τ) for ALS-033719 and ALS-033927, oseltamivir, oseltamivir carboxylate, and JNJ-63623872 | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on days 7, 8, and 14 for ALS-033719, ALS-033927, and JNJ-63623872
Area under plasma concentration-time curve from time 0 to last measurable plasma concentration (AUClast) for digoxin, midazolam 1'-OH-midazolam, and pitavastatin | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on Days 1, 11, and 17 for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin
Maximum observed plasma concentration (Cmax) for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on Days 1, 11, and 17 for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin

SECONDARY OUTCOMES:
Last observed plasma concentration (Clast) for ALS-033719, ALS-033927, oseltamivir, oseltamivir carboxylate, JNJ-63623872, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin when applicable | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on days 7, 8, and 14 for ALS-033719, ALS-033927, and JNJ-63623872, Days 1, 11, and 17 for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin
Terminal elimination half-life (t½) for ALS-033719, ALS-033927, oseltamivir, oseltamivir carboxylate, JNJ-63623872, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin when applicable | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on days 7, 8, and 14 for ALS-033719, ALS-033927, and JNJ-63623872, Days 1, 11, and 17 for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin
Time of the maximum observed plasma concentration (tmax) for ALS-033719, ALS-033927, oseltamivir, oseltamivir carboxylate, JNJ-63623872, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin when applicable | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on days 7, 8, and 14 for ALS-033719, ALS-033927, and JNJ-63623872, Days 1, 11, and 17 for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin
Time to last measurable plasma concentration (tlast) for ALS-033719, ALS-033927, oseltamivir, oseltamivir carboxylate, JNJ-63623872, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin when applicable | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on days 7, 8, and 14 for ALS-033719, ALS-033927, and JNJ-63623872, Days 1, 11, and 17 for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin
Apparent oral clearance (CL/F) for ALS-033719, ALS-033927, oseltamivir, oseltamivir carboxylate, JNJ-63623872, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin when applicable | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on days 7, 8, and 14 for ALS-033719, ALS-033927, and JNJ-63623872, Days 1, 11, and 17 for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin
Apparent volume of distribution (Vz/F) for ALS-033719, ALS-033927, oseltamivir, oseltamivir carboxylate, JNJ-63623872, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin when applicable | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on days 7, 8, and 14 for ALS-033719, ALS-033927, and JNJ-63623872, Days 1, 11, and 17 for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin
Apparent terminal elimination rate constant (λz) for ALS-033719, ALS-033927, oseltamivir, oseltamivir carboxylate, JNJ-63623872, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin when applicable | At 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose on days 7, 8, and 14 for ALS-033719, ALS-033927, and JNJ-63623872, Days 1, 11, and 17 for oseltamivir, oseltamivir carboxylate, digoxin, midazolam, 1'-OHmidazolam, and pitavastatin
Number of participants with treatment emergent adverse events | From Day 1 to Day 29
Change from baseline in 4β-hydroxycholesterol (Group 3 only) | From Day 1 to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom